CLINICAL TRIAL: NCT01310426
Title: Risk Factors for Anal Sphincter Damage During Vaginal Delivery
Acronym: AnaSphRF
Status: Completed | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: AnaSphRF-HMO-CTIL
Record Dates: First submitted 2011-03-01; First posted 2011-03-08 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Anal Sphincter Injury; Fecal Incontinence
Keywords: Anal Sphincter injury; Fecal Incontinence
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- anal sphincter damage: After assessing women after vaginal delivery, a comparison will be made between those with anal sphincter damage and those women without.
  Interventions: Other: 3D transperineal Ultrasound

INTERVENTIONS:
Other: 3D transperineal Ultrasound — 3D transperineal Ultrasound after vaginal delivery

SUMMARY:
Vaginal delivery may cause various levels of damage to the anal sphincter. According to the literature, one third - two third of women diagnosed with 3rd degree rupture during vaginal delivery suffer from fecal incontinence. This has an adverse effect on the quality of life. Different risk factors such as: first births, instrumental delivery, high birth weight, prolonged second stage, epidural anesthesia etc. were assessed and found to be associated with anal sphincter disruption. The purpose of this study is to assess risk factors for anal sphincter disruption by new methods such as three-Dimensional transperineal ultrasound (3D transperineal US).

ELIGIBILITY:
Inclusion Criteria:

* First Delivery
* Vaginal Delivery
* Birthweight > 3000
* Singleton pregnancy

Exclusion Criteria:

* Anal sphincter disruption before birth

Ages: 17 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study population are women between ages 17 and 40 after their first delivery at the Hadassa Mount Scopus hospital in Jerusalem, Israel.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2011-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Anal sphincter damage | up to one year after vaginal birth
  Anal Sphincter Damage wil be assessed by usin 3D transperineal US in women after vaginal delivery

CONTACTS AND LOCATIONS:
Overall Officials: Drorith Hochner, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel